CLINICAL TRIAL: NCT01657240
Title: Phase 3 Clinical Trial to Evaluate the Clinical Efficacy of PRO-118 Compared With Olopatadine Hydrochloride Ophthalmic Solution in Allergic Conjunctivitis
Brief Title: Clinical Efficacy of PRO-118 Compared With Olopatadine Hydrochloride Ophthalmic Solution in Allergic Conjunctivitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Formula Reformulation
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH118-0112/III
Record Dates: First submitted 2012-07-19; First posted 2012-08-06 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO-118 (Experimental): pro-118 ophthalmic solution, instill one drop in each eye once a day for 21 days
  Interventions: Drug: PRO-118
- Olopatadine Hydrochloride (Active Comparator): Olopatadine Hydrochloride ophthalmic solution 2%, instill one drop in each eye once a day for 21 days
  Interventions: Drug: Olopatadine Hydrochloride

INTERVENTIONS:
Drug: PRO-118 — instill one drop in each eye once a day for 21 days
  Other Names: PRO-118 ophthalmic solution
  Arms: PRO-118
Drug: Olopatadine Hydrochloride — instill one drop in each eye once a day for 21 days
  Other Names: Olopatadine Hydrochloride ophthalmic solution
  Arms: Olopatadine Hydrochloride

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of the ophthalmic solution PRO-118 compared with olopatadine hydrochloride ophthalmic solution in allergic conjunctivitis.

DETAILED DESCRIPTION:
Allergic conjunctivitis is inflammation of the tissue lining the eyelids (conjunctiva) due to a reaction from allergy-causing substances. The main aim in allergic conjunctivitis is to improve the quality of life in these patients. Antihistaminic medication is commonly used to treat allergic conjunctivitis symptoms. The aim of the study is to compare the clinical efficacy of two ophthalmic solutions containing each one an antihistaminic drug.

A phase III randomized double-blind clinical trial will be conducted to evaluate efficacy of the ophthalmic solution PRO-118 compared with olopatadine hydrochloride ophthalmic solution in allergic conjunctivitis. Patients will be randomized to receive one of the treatments for 21 days. Efficacy endpoints will be measured at baseline and at 21 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Allergic conjunctivitis diagnosis
* Both genders
* Age between 6 and 60 years
* Patients with no treatment 2 years prior to study inclusion

Exclusion Criteria:

* Patients with one blind eye
* Visual acuity < 20/40 in any eye
* Patients with any active ocular disease that would interfere with study interpretation
* Patients in treatment with any medication that could interfere with the study, contraindication of any medication used in the protocol
* Patients with: diabetes mellitus, rheumatoid arthritis, hypertension, or any type of cancer
* Patients with history of hypersensitivity or contraindication for any drug used in the study
* Patients receiving systemic or topical treatment based on antihistamines, corticosteroids or immunomodulators
* Pregnant patients, at risk of pregnancy or breastfeeding
* Patients without birth control treatment
* Patients who had participated in any clinical trial in the last 90 days

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
conjunctival hyperemia | day 21
  Change from Baseline in conjunctival hyperemia after 21 days of treatment

SECONDARY OUTCOMES:
epiphora | day 21
  Change from Baseline in epiphora after 21 days of treatment

OTHER OUTCOMES:
green lissamine dye | day 21
  Number of patients with normal green lissamine dye
fluorescein dye | day 21
  Number of patients with normal fluorescein dye